CLINICAL TRIAL: NCT05083624
Title: Feasibility and Prognosis of Early Rehabilitation in Patients With Extracorporeal Membrane Oxygenation
Brief Title: Feasibility and Prognosis of Early Rehabilitation in Patients With ECMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JinyanXing (Other)
Responsible Party: Sponsor-Investigator, JinyanXing, Director, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: QYFYKYLL9121011920
Record Dates: First submitted 2021-09-30; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Extracorporeal Membrane Oxygenation
Keywords: Extracorporeal Membrane Oxygenation; early rehabilation; muscle ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation group (Experimental)
  Interventions: Behavioral: rehabilation therapy
- control group (No Intervention): adhere to standardized management guidelines for anticoagulation, ventilation, sedation specific to the MICU ECMO population

INTERVENTIONS:
Behavioral: rehabilation therapy — After comprehensive assessment by doctors, nurses and rehabilitation therapists, patients gradually begin rehabilitation treatment.IMS 0: no mobilisation or passively exercised by staff. IMS 1: sitting in bed and actively exercising .IMS 2: passively moved to chair without standing.IMS 3: sitting over edge of bed.IMS 4: standing in front of bed.IMS 5: transferring bed to chair.IMS 6: marching on spot.IMS 7: walking with assistance of more than one person.IMS 8: walking with assistance of one person.IMS 9: walking independently with a gait aid.IMS 10: walking independently without a gait aid.
  Arms: Rehabilitation group

SUMMARY:
ECMO is increasingly used in critically ill patients with severe circulatory and/or respiratory failure. Because of the catheterization of the femoral artery and femoral vein, usage of sedatives, and occasionally with neuromuscular blockers, ECMO patients are generally considered unsuitable for early activity. However, some recent retrospective studies and a small number of single-center, small-scale prospective studies have shown that early activity of ECMO patients is feasible, and early active activity is associated with recovery of independent function and reduction of delirium incidence.

ELIGIBILITY:
Inclusion Criteria:

* ECMO time ≥1 day
* Aged older than16 years old and less than 70 years old

Exclusion Criteria:

* coma deep
* sedation muscle relaxation (RAAS-3-5)
* Active bleeding deep vein thrombosis
* High dose of vasoactive drugs
* unstable vital signs
* Acute stage of myocardial infarction (within 2d)
* Malignant arrhythmia
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
muscle ultrasound | 7 days
  The thickness of intercostal muscle and rectus femoris muscle was measured by ultrasound

SECONDARY OUTCOMES:
ECMO duration time | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided